CLINICAL TRIAL: NCT02284308
Title: ELDAPT: Elderly With Locally Advanced Lung Cancer: Deciding Through Geriatric Assessment on the oPtimal Treatment Strategy
Brief Title: Elderly With Locally Advanced Lung Cancer: Deciding Through Geriatric Assessment on the Optimal Treatment Strategy
Acronym: ELDAPT
Status: Active, not recruiting | Type: Observational
Sponsor: Maastricht Radiation Oncology (Other)
Collaborators: Dutch Society of Physicians for Pulmonology and Tuberculosis (Other); Erasmus Medical Center (Other); VieCuri Medical Centre (Other); AstraZeneca (Industry); Dutch Cancer Society (Other)
Responsible Party: Sponsor
Other Study IDs: ELDAPT
Record Dates: First submitted 2014-10-30; First posted 2014-11-06 (Estimated); Last update posted 2025-07-04 (Actual); Status verified 2025-07

CONDITIONS: NSCLC
Keywords: NSCLC

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Patients with any subtype of NSCLC, primary UICC Stage III, age ≥ 75 years: All registered patients will undergo a geriatric assessment to assess vulnerability. Based on this assessment, patients are offered treatment according to the discretion of the physician and patient.

SUMMARY:
There is no detailed information available on benefits and harms of intensified treatment with concurrent RCHT among a subpopulation of elderly patients. Reliable tools are needed to distinguish the subgroup of fit patients from frail patients.

DETAILED DESCRIPTION:
Lung cancer is a problem of the elderly: 30% of the lung cancer patients are aged ≥ 75 years. Due to underrepresentation of elderly patients in clinical trials there is a lack of evidence to select the optimal treatment strategy for these patients. Concurrent radiochemotherapy (RCHT) has been recognised as the standard treatment of stage III NSCLC patients with a good performance status. Evidence for this treatment was gained in clinical trials that mostly excluded elderly patients. Furthermore, the survival gain obtained with combined RCHT, comes with a significant increase in toxicity. Therefore, information on benefits and harms of intensified treatment with concurrent RCHT among a subpopulation of medically fit elderly patients is still lacking. Moreover, reliable tools are needed to distinguish the subgroup of fit patients from frail patients, i.e. those expected to experience important toxicity.

ELIGIBILITY:
Inclusion criteria (according to the protocol):

* Any subtype of pathologically proven NSCLC, primary UICC Stage III disease;
* Age ≥ 75 years;
* No surgery or adjuvant chemotherapy for NSCLC in the last year;
* No prior radiotherapy to the ipsilateral thorax or mediastinum;
* No clinical superior vena cava syndrome;
* No diagnosis of other cancer within the last 3-years (except in situ carcinoma's and / or non-melanoma skin cancer);
* Written informed consent

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Patients aged ≥ 75 years, with any subtype of NSCLC, stage III
Sampling Method: Non-Probability Sample
Enrollment: 180 (Actual)
Dates: Start 2016-07 (Actual); Primary Completion 2025-01-01 (Actual); Study Completion 2029-12-18 (Estimated)

PRIMARY OUTCOMES:
Correlation GA with QAS (quality adjusted survival) | 5 years
  To corellate results of the geriatric assessment with quality-adjusted survival (QAS) after radical intent therapy in patients with stage III NSCLC ≥75 years

SECONDARY OUTCOMES:
Geriatric assessment | Baseline
  To perform a geriatric assessment in stage III NSCLC patients to distinguish patients fit enough to undergo intensified treatment and to develop a reliable and clinically applicable geriatric screening instrument to guide treatment decisions in stage III NSCLC
Medical comparison between treatments | 5 years
  To compare different treatment strategies for fit elderly patients with respect to overall and quality adjusted survival
Cost-effectiveness | End of study
  To compare cost-effectiveness of sequential and concurrent RCHT for fit elderly patients with stage III NSCLC
Development and validation of geriatric screening instrument | 5 years
  To develop and validate a clinically applicable geriatric screening instrument that enables appropriate treatment stratification in the elderly NSCLC patient
Flow chart | 5 years
  To develop a flow chart for cost-effective clinical decision-making, in clinical practice
Predictive value | 5 years
  To determine the predictive value of saliva biomarkers on QAS in elderly patients with stage III NSCLC

CONTACTS AND LOCATIONS:
Overall Officials: Judith van Loon, MD, PhD, Principal Investigator — Maastro (radiotherapist); Anne-Marie Dingemans, MD, PhD, Principal Investigator — Erasmus Medical Center; Mariska Janssen-Heijnen, PhD, Principal Investigator — VieCuri Medical Centre
Locations (22):
- Netherlands (22):
  - Ziekenhuisgroep Twente, Almelo
  - Gelre ziekenhuis, Apeldoorn
  - Radiotherapiegroep Arnhem, Arnhem
  - Rijnstate, Arnhem
  - Deventer Hospital, Deventer
  - Gelderse Vallei, Ede
  - Catharina Ziekenhuis, Eindhoven
  - Máxima MC, Eindhoven
  - Medisch Spectrum Twente, Enschede
  - Rivas Zorggroep, Gorinchem
  - Groen Hart Ziekenhuis, Gouda
  - Zuyderland, Heerlen
  - Maastro, Maastricht
  - MUMC+, Maastricht
  - Canisius-Wilhelmina Hospital, Nijmegen
  - Laurentius Hospital, Roermond
  - Maasstad Ziekenhuis, Rotterdam
  - Ikazia Ziekenhuis, Rotterdam
  - Haga Ziekenhuis, The Hague
  - Haaglanden MC, The Hague
  - VieCuri MC, Venlo
  - Zaans MC, Zaandam

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Driessen EJM, van Loon JGM, Maas HA, Dingemans AC, Janssen-Heijnen MLG. Geriatric Assessment for Older Patients with Non-small Cell Lung Cancer: Daily Practice of Centers Participating in the NVALT25-ELDAPT Trial. Lung. 2018 Aug;196(4):463-468. doi: 10.1007/s00408-018-0116-8. Epub 2018 Apr 12. PMID 29651598